CLINICAL TRIAL: NCT01061294
Title: Evaluation of Outcomes Using the AMO Advanced Customvue™ iLasik Procedure (Wavescan Wavefront® System, Star S4 IR™ Excimer Laser System and Intralse™ FS System)
Brief Title: Evaluation of Outcomes Using the AMO Advanced Customvue™ iLasik Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: William Trattler, The Center for Excellence in Eye Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iLASIK
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Vision Correction
Keywords: Assess the efficacy, predictability and safety of the Advanced CustomVue™ iLASIK procedure.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced CustomVue™ iLASIK procedure (Other)
  Interventions: Procedure: Advanced CustomVue™ iLASIK procedure; Device: WaveScan WaveFront® System, STAR S4 IR™ Excimer Laser System and IntraLase™ FS System

INTERVENTIONS:
Procedure: Advanced CustomVue™ iLASIK procedure
Device: WaveScan WaveFront® System, STAR S4 IR™ Excimer Laser System and IntraLase™ FS System

SUMMARY:
The purpose of this study is to assess the efficacy, predictability and safety of the Advanced CustomVue™ iLASIK procedure (WaveScan WaveFront® System, STAR S4 IR™ Excimer Laser System and IntraLase™ FS System). Patient data will be collected electronically and analyzed to determine improvements in postoperative visual acuity, visual quality and residual error.

ELIGIBILITY:
Inclusion Criteria:

1. the subject must be male or female, of any race, and at least 21 years old at the time of the pre-operative examination;
2. both eyes must have a BSCVA of 20/20 or better;
3. both eyes must have a manifest refractive error from -0.50 D to -6.00 D, a cylinder component up to -3.00 D, and a maximum manifest spherical equivalent of -6.00 D;
4. both eyes must have a minimum pupil size of at least 6.0mm in dim illumination on wavescan;
5. both eyes must demonstrate refractive stability confirmed by clinical records or previous glasses. Refractive stability shall be documented by a change of less than or equal to 0.50 diopter (sphere and cylinder) at an exam at least 12 months prior to the baseline examination. The astigmatic axis must also be within 15 degrees for eyes with cylinder greater than 0.50 D; and
6. subjects should be willing and capable of returning for follow-up examinations for the duration of the study.

Exclusion Criteria:

1. subjects who use concurrent topical or systemic medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment; NOTE: The use of topical or systemic corticosteroids, whether chronic or acute, is deemed to adversely affect healing and subjects using such medication are specifically excluded from eligibility.
2. subjects with a history of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis; NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, will specifically exclude subjects from eligibility.
3. the subject must not have a history of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or with evidence of glaucoma or propensity for narrow angle glaucoma in either eye; NOTE: This includes any subject with open angle glaucoma, regardless of medication regimen or control. .
4. the subject must not have any evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye;
5. subjects with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course;
6. patients who do not achieve Iris registration at the time of their wavescan; and
7. patients seeking monovision.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative visit procedures will include visual acuity and quality assessments and monitoring for surgical complications necessitating retreatment. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- William Trattler, Miami, Florida, United States